CLINICAL TRIAL: NCT06960798
Title: Characterizing the Genomic Landscape of Prostate Cancer in Native American Populations (Nat-Geno)
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-NAT-Geno
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Native American Men; Genomic Profile
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archived tumor tissue collected at screening.
  Blood samples collected within the first year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Native American Group: 150 patients will be assigned in this group.
  Interventions: Other: Bio-specimen Collection; Other: Blood Draw

INTERVENTIONS:
Other: Bio-specimen Collection — Tissue samples will be taken from existing archived collections and sent for further analysis.
Other: Blood Draw — Blood samples will be collected within the first year of enrollment.

SUMMARY:
The purpose of this study is to analyze tumor tissue samples from patients of Native American identity with prostate cancer. By examining these samples, researchers hope to understand how different genes in your tumor can influence treatment decisions, how your cancer progresses and the outcome of your cancer.

DETAILED DESCRIPTION:
This study aims to establish a comprehensive database of Native American (NA) patients diagnosed with prostate cancer (PC), focusing on an in-depth characterization of the genomic landscape. Archived tumor tissue collected at screening and peripheral blood samples obtained within the first year of enrollment will serve as the basis for comprehensive molecular analyses. Whole exome sequencing (WES) and whole transcriptome sequencing (RNA-seq) will be performed to characterize and delineate the genomic and transcriptomic landscape of the study cohort. The study will initially enroll participants at the Stephenson Cancer Center, with planned expansion to additional sites across Oklahoma and, subsequently, to other institutions across the United States. Oversight will be maintained by the Tribal Institutional Review Board and an independent Community Advisory Board to ensure cultural appropriateness, transparency, and sustained community engagement throughout the research process. The overarching objective is to generate insights that will inform the development of personalized treatment strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by the patient prior to the performance of any study-specific procedures, sampling, or analyses.
* At least 18 years-of-age at the time of signature of the informed consent form (ICF).
* Patients who self-identify as Native American.
* Patients with a pathologically proven diagnosis of PC (any stage).
* Availability of most recent archived tumor samples.

Exclusion Criteria:

* Patients not of Native American descent or identity.
* Patient does not have archival tissue available.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be male due to the type of cancer being observed it is not prevalent in females.
Study Population: This clinical trial will focus on addressing the underrepresented Native American population served by the Urology Oncology Department at Stephenson Cancer Center. To broaden the scope of data, the trial will also involve other institutions, while maintaining its primary focus on the target population.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-05-02 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in the genomic profiles of Prostate Cancer | 1-3 years
  Comprehensively characterize the genomic profile of prostate cancer in Native American patients compared to Caucasian patients. Genetic testing will be conducted using Caris Whole Exome Sequencing (WES) and Whole Transcriptome Sequencing (WTS).

SECONDARY OUTCOMES:
Comparison of Genomic Profiles | 1-3 years
  The study compares the Native American population with a reference Caucasian cohort to characterize molecular disparities and evaluate their clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Adanma Ayanambakkam, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No